CLINICAL TRIAL: NCT04910347
Title: A Phase 2, Open-label Trial of Consolidation Nivolumab After Concurrent Chemoradiotherapy in Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Consolidation Nivolumab After Concurrent Chemoradiotherapy in Locally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Chang Gon Kim, Principal Investigator, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-0330
Record Dates: First submitted 2021-05-18; First posted 2021-06-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Nivolumab
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Dosage within 12 weeks after the end of concurrent chemoradiation therapy. Nivolumab 360mg Intravenously administered every 3 weeks.
  As a consolidation regimen, administration of Nivolumab is administered for up to a total of 1 year until disease progression or unacceptable to toxicity occurs.

SUMMARY:
The clinical efficacy of nivolumab for locally advanced nasopharyngeal carcinoma patients with residual disease after standard chemoradiotherapy is not known. In this study, we aim to investigate the role of nivolumab in locally advanced NPC after chemoradiotherapy the safety profile and antitumor activity of the anti-programmed death 1 (PD-1) receptor monoclonal antibody, nivolumab after in patients with advanced nasopharyngeal carcinoma

DETAILED DESCRIPTION:
Dosage within 12 weeks after the end of concurrent chemoradiation therapy. Nivolumab 360mg Intravenously administered every 3 weeks.

As a consolidation regimen, administration of Nivolumab is administered for up to a total of 1 year until disease progression or unacceptable to toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age (at the time of informed consent): 19 years and older
3. Subjects with histologically- or cytologically-confirmed advanced Nasopharyngeal cancer (Stage II -IVa) according to 8th edition clinical staging system of the American Joint Committee on Cancer before the start of concurrent chemoradiotherapy
4. Patients who have recovered from previous toxicities of standard chemoradiotherapy (Grade ≤1).
5. ECOG (Eastern Cooperative Oncology Group) Performance Status Score 0 or 1
6. Patients with a life expectancy of at least 3 months
7. Patients whose latest laboratory data meet the below criteria within 7 days before registration. If the date of the laboratory tests at the time of registration is not within 7 days before the first dose of the investigational product, testing must be repeated within 7 days before the first dose of the investigational product, and these latest laboratory tests must meet the following criteria. Of note, laboratory data will not be valid if the patient has received a granulocyte colony-stimulating factor (G-CSF) or blood transfusion within 14 days before testing.

   * White blood cells ≥2,000/mm3 and neutrophils ≥1,500/mm3
   * Platelets ≥100,000/mm3
   * Hemoglobin ≥9.0 g/dL
   * AST (GOT) and ALT (GPT) ≤3.0-fold the upper limit of normal (ULN) of the study site (or ≤5.0-fold the ULN of the study site in patients with liver metastases)
   * Total bilirubin ≤1.5-fold the ULN of the study site
   * Creatinine ≤1.5-fold the ULN of the study site or creatinine clearance (either the measured or estimated value using the Cockcroft-Gault equation) >45 mL/min
8. Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons) #1 must agree to use contraception#2 from the time of informed consent until 5 months or more after the last dose of the investigational product. Also, women must agree not to breastfeed from the time of informed consent until 5 months or more after the last dose of the investigational product.
9. Men must agree to use contraception#2 from the start of study treatment until 7 months or more after the last dose of the investigational product.

   * Women of childbearing potential are defined as all women after the onset of menstruation who are not postmenopausal and have not been surgically sterilized (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy). Postmenopause is defined as amenorrhea for ≥12 consecutive months without specific reasons. Women using oral contraceptives, intrauterine devices, or mechanical contraception such as contraceptive barriers are regarded as having childbearing potential.
   * The subject must consent to use any two of the following methods of contraception: vasectomy or condom for patients who are male or female subject's partner and tubal ligation, contraceptive diaphragm, intrauterine device, spermicide, or oral contraceptive for patients who are female or male subject's partner.

Exclusion Criteria:

1. Patients with multiple primary cancers (with the exception of completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, or superficial bladder cancer, or any other cancer that has not recurred for at least 5 years)
2. Patients with residual adverse effects of prior therapy or effects of surgery that would affect the safety evaluation of the investigational product in the opinion of the investigator or sub-investigator.
3. Patients with current or past history of severe hypersensitivity to any other antibody products
4. Patients with concurrent autoimmune disease or history of chronic or recurrent autoimmune disease
5. Patients with a current or past history of interstitial lung disease or pulmonary fibrosis diagnosed based on imaging or clinical findings. Patients with radiation pneumonitis may be randomized if the radiation pneumonitis has been confirmed as stable (beyond acute phase) without any concerns about recurrence.
6. Patients with concurrent diverticulitis or symptomatic gastrointestinal ulcerative disease
7. Patients with any metastasis in the brain or meninx that is symptomatic or requires treatment. Patients may be randomized if the metastasis is asymptomatic and requires no treatment.
8. Patients with pericardial fluid, pleural effusion, or ascites requiring treatment
9. Patients with uncontrollable, tumor-related pain
10. Patients who have experienced a transient ischemic attack, cerebrovascular accident, thrombosis, or thromboembolism (pulmonary arterial embolism or deep vein thrombosis) within 180 days before registration
11. Patients with a history of uncontrollable or significant cardiovascular disease meeting any of the following criteria:

    * Myocardial infarction within 180 days before registration
    * Uncontrollable angina pectoris within 180 days before registration
    * New York Heart Association (NYHA) Class III or IV congestive heart failure
    * Uncontrollable hypertension despite appropriate treatment (e.g., systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥ 90 mmHg lasting 24 hours or more)
    * Arrhythmia requiring treatment
12. Patients receiving or requiring anticoagulant therapy for a disease. Patients receiving antiplatelet therapy including low-dose aspirin may be enrolled.
13. Patients with uncontrollable diabetes mellitus
14. Patients with systemic infections requiring treatment
15. Patients who have received systemic corticosteroids (except for temporary use, e.g., for examination or prophylaxis of allergic reactions) or immunosuppressants within 28 days before registration
16. Patients who have received antineoplastic drugs (e.g., chemotherapy agents, molecular-targeted therapy agents, or immunotherapy agents) within 28 days before registration
17. Patients who have undergone surgical adhesion of the pleura or pericardium within 28 days before registration
18. Patients who have undergone surgery under general anesthesia within 28 days before registration
19. Patients who have undergone surgery involving local or topical anesthesia within 14 days before registration
20. Patients who have received radiotherapy within 28 days before registration, or radiotherapy to bone metastases within 14 days before registration
21. Patients who have received any radiopharmaceuticals (except for examination or diagnostic use of radiopharmaceuticals) within 56 days before registration
22. Patients with a positive test result for any of the following: HIV-1 antibody, HIV-2 antibody, HTLV-1 antibody, HBs antigen, or HCV antibody (except if HCV-RNA negative)
23. Patients with a negative HBs antigen test but a positive test result for either HBs antibody or HBc antibody with a detectable level of HBV-DNA
24. Women who are pregnant or breastfeeding, or possibly pregnant
25. Patients who have received any other unapproved drug (e.g., investigational use of drugs, unapproved combined formulations, or unapproved dosage forms) within 28 days before registration
26. Patients who have previously received Nivolumab, anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, anti-CD137 antibody, anti-CTLA-4 antibody or other therapeutic antibodies or pharmacotherapies for regulation of T-cells
27. Patients judged to be incapable of providing consent for reasons such as concurrent dementia
28. Other patients judged by the investigator or sub-investigator to be inappropriate as subjects of this study
29. Patient with current or past history of hypersensitivity to Nivolumab.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 2years | 2 years
  Progression-free survival rate at 2 years, which is the primary endpoint, will be measured by the proportion of patients who remain progression-free after 2 years of study registration.

SECONDARY OUTCOMES:
Object response rate (ORR) | Screening, Every 3months during the administration period(up to 1year), every 6 months after the end of the administration(up to 5years)
  according to RECIST 1.1 criteria
Overall survival (OS) | Intervals of 6 months up to 5 years after the end of dosing
  Overall survival will be followed continuously while subjects are on the study drug and every 6 months after discontinuation or progression for up to 5 years following the start of therapy either by direct contact (office visits) or via telephone contact, until death, withdrawal of study consent, or lost to follow-up.
Subject with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | Every cycle (every 3weeks), until 28 days after the end of treatment.
  The procedures and assessments may be performed as part of standard of care; however, data for these assessments should remain in the subject's medical record and should not be provided to Ono unless specifically requested. NCI CTCAE Version 5.0 will be the criteria used to assess adverse events.
Multiplexed biomarker analysis of tumor and immune cells in the TME | At screening, At cycle2 day1(each cycle is 28 days), End of treatment (up to a total of 1 year)
  To understand correlated expressions of protein markers related to therapy response, multiplexed-image analysis (Vectra Polaris® and inForm®, PerkinElmer) is applied in tumor tissues
Analysis of gene expression profile and immune markers | At screening, At cycle2 day1(each cycle is 28 days), End of treatment (up to a total of 1 year)
  Analysis of gene expression profile and immune markers with tissue and peripheral blood
Soluble factor analysis | At screening, At cycle2 day1(each cycle is 28 days), End of treatment (up to a total of 1 year)
  Soluble factor analysis with blood: Cytokines related to adaptive immune responses, chemokines, and VEGF will be analyzed using the Cytometric Bead Assay (CBA) from serially collected plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Hye Ryun Kim, Principal Investigator — Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No